CLINICAL TRIAL: NCT05352581
Title: Clinical Evaluation of The BD Veritor™ At-Home COVID-19 & Flu Test and BD Veritor™ System for Rapid Detection of SARS-CoV-2 & Flu A+B Assay
Brief Title: BD Veritor™ At-Home and BD Veritor™ Professional
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: IDS-VERTPPGEN2
Record Dates: First submitted 2022-04-11; First posted 2022-04-29 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Upper Respiratory Infection
Keywords: SARS COV 2; Influenza
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Self-collected and clinician collected nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- BD Veritor: Each subject will:
  Self collect a nasal swab for testing on the BD Veritor At-home test (test device) Have a clinician collected nasal swab for testing on the BD Veritor Professional Test (test device) Have a clinical collected nasal swab for testing on an FDA cleared/approved RT-PCR assay (control device)
  Interventions: Diagnostic Test: BD Veritor At-Home; Diagnostic Test: BD Veritor Professional

INTERVENTIONS:
Diagnostic Test: BD Veritor At-Home — BD Veritor At-Home rapid self testing
Diagnostic Test: BD Veritor Professional — BD Veritor Professional rapid test

SUMMARY:
The BD Veritor™ System is a rapid test that is testing for both COVID-19 and for Influenza This study will try to determine if the BD Veritor™ system can assist in the diagnosis of someone who has upper respiratory infection symptoms. There is both an At-Home self test and test completed by a health care professional that will be completed during this study.

DETAILED DESCRIPTION:
This is a prospective, multi-country, multicenter, comparative study to assess the performance of the BD Veritor™ At-Home SARS-CoV-2 & Flu A+B test and the BD Veritor™ System for Rapid Detection of SARS-CoV-2 & Flu A+B (Professional use) compared to an FDA approved Flu A/B reference assay (RT-PCR) and FDA authorized molecular SARS-CoV-2 comparator reference method assays.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants symptomatic of an acute respiratory illness within 7 DOSO
* 2. ≥2 years of age at the time of study participation
* 3. Symptomatic subjects with
* a. Any one of the following symptoms (with or without additional symptoms):
* i. Fever
* 1. Oral/temporal artery: ≥100.4 °F / ≥38.0 °C
* 2. Rectal/Ear: ≥101.2 °F / ≥38.5 °C
* ii. Cough
* iii. Malaise (fatigue/extreme tiredness)
* b. Or two of the following symptoms:
* i. Sore throat,
* ii. Shortness of breath/difficult breathing
* iii. Rhinorrhea (runny or stuffy nose),
* iv. Myalgia,
* v. Headache,
* vi. Sneezing,
* vii. New loss of taste or smell,
* viii. One or more GI symptoms (nausea, vomiting, diarrhea)

Exclusion Criteria:

* 1. Participants currently undergoing treatment and/or within the past thirty (30) days of the study, with medication to treat novel Coronavirus SARS-CoV-2 viral infections, which may include but is not limited to Remdesivir (Veklury)
* 2. Participants receiving convalescent plasma therapy for SARS-CoV-2.
* 3. Participants who have received antiviral medications for influenza within the previous 30 days.
* 4. Participants who have had a nasal wash or aspirate as part of their standard of care treatment on day of study visit.
* 5. The participant is currently receiving or has received within the past thirty (30) days of the study visit, an experimental biologic or drug including either treatment or therapy.
* 6. Participants who have been previously enrolled in the study.
* 7. History of frequent or difficult to control nosebleeds within the last fourteen (14) days.
* 8. Participants who have tested positive for Flu A/B or SARS-CoV-2 within the last 28 days (excluding the day of enrollment in the study).

Exclusion criteria for the participation in the At-Home portion of the study would include all of the criteria previously listed and include the following

* 1. Participants without the ability to read or write in the English Language
* 2. Participants with prior medical or laboratory training.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals presenting with symptoms of acute respiratory illness
Sampling Method: Non-Probability Sample
Enrollment: 1146 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the BD Veritor At-Home Assay | Immediately after specimen collection
  Positive percent agreement of the BD Veritor At-Home Assay compared to an FDA cleared/approved RT-PCR Assay
Diagnostic accuracy of the BD Veritor Professional Assay | Immediately after specimen collection
  Positive percent agreement of the BD Professional Assay compared to an FDA cleared/approved RT-PCR Assay

SECONDARY OUTCOMES:
Ease of Use of the BD Veritor At-Home Assay | Within 30 minutes of test completion
  Subject completed 5-Point Likert scale rating ease of use where 1 indicates difficult and 5 indicates easy
Ease of Use of the BD Professional Assay | Within 1 day of first device use
  Clinician completed 5-Point Likert scale rating ease of use where 1 indicates difficult and 5 indicates easy

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - CTMD Research, Coconut Creek, Florida
  - CTMD Research, Palm Springs, Florida
  - DBC Research, Pembroke Pines, Florida
  - CTMD Reserarch, Asheville, North Carolina
  - Kur Research - AFC Urgent Care, Easley, South Carolina
  - Kur Research - AFC Urgent Care, Powdersville, South Carolina
  - Kur Research - AFC Urgent Care, Seneca, South Carolina
  - Kur Research - Complete Health Partners, Hendersonville, Tennessee
  - Kur Research - Complete Health Partners, Nashville, Tennessee
- University of the Sunshine Coast, Sippy Downs, Queensland, Australia
- New Zealand (7):
  - Southern Clinical Trials - Totara, Auckland
  - Optimal Clinical Trials, Auckland
  - Southern Clinical Trials - Remuera, Auckland
  - Lakeland Clinical Trials - Waikato, Hamilton
  - Southern Clinical Trials - Tasman, Nelson
  - Silverdale Medical Ltd, Silverdale
  - Southern Clinical Trials - Wellington, Upper Hutt